CLINICAL TRIAL: NCT02864355
Title: Does Perioperative Goal Directed Therapy Using Flotrac Improve Outcomes in Esophagectomy Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Minimally invasive surgical methods have ceased enrollment
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00045623
Record Dates: First submitted 2016-07-15; First posted 2016-08-12 (Estimated); Results first posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Early Goal-Directed Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Goal Directed Therapy (Active Comparator): In this arm patient will have the FloTrac monitor and a Goal Directed Therapy algorithm will be used to manage blood pressures.
  Interventions: Device: Goal Directed Therapy
- Usual Care (No Intervention): Standard of care will be used to manage blood pressures.

INTERVENTIONS:
Device: Goal Directed Therapy — Participants in this group will have a FloTrac monitor attached to their arterial line and the Goal Directed Therapy algorithm will be followed to manage blood pressures.
  Arms: Goal Directed Therapy

SUMMARY:
The objective of this prospective, randomized controlled study is to ascertain whether the perioperative use of the FloTrac device to guide fluid and vasopressor management during esophagectomy improves patient outcomes. The primary outcome is cardiopulmonary complications; however, the secondary outcome of decreasing patient morbidity (acute renal injury, anastomotic leak, and overall length of both ICU (intensive care unit) and hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Patients undergoing primary resection of esophageal cancer and resultant esophagectomy.

Exclusion Criteria:

* Patients < 55kg or > 140 kg, based on literature regarding accuracy of FloTrac.
* Patients with sustained preoperative dysrhythmias, based on literature regarding accuracy of FloTrac (atrial flutter and/or atrial fibrillation).
* Patients with diagnosed NYHA class III-IV failure or documented EF < 30%
* Patients who are unable/unwilling to consent for study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-06; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Guldan, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was stopped early due to to insufficient enrollment accruals
Period: Overall Study
Arm/Group | Goal Directed Therapy | Usual Care
Started | 25 | 28
Completed | 23 | 25
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Goal Directed Therapy | Usual Care | Total
Number analyzed (Participants) | 23 | 25 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 12 | 22
  >=65 years | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (8.8) | 62.8 (15.2) | 63.9 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 16 | 17 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 19 | 23 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 25 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cardiopulmonary Complications
Description: Any documented cardiopulmonary complications present upon chart review.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Goal Directed Therapy | Usual Care
Number analyzed (Participants) | 23 | 25
Participants | 8 | 11

2. Secondary Outcome: Anastomotic Leak Diagnosed Via Radiograph
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Goal Directed Therapy | Usual Care
Number analyzed (Participants) | 23 | 25
Participants | 1 | 1

3. Secondary Outcome: Number of Participants With Renal Injury
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Goal Directed Therapy | Usual Care
Number analyzed (Participants) | 23 | 25
Participants | 3 | 3

4. Secondary Outcome: Death
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Goal Directed Therapy | Usual Care
Number analyzed (Participants) | 23 | 25
Participants | 2 | 1

5. Secondary Outcome: Length of Intensive Care Unit Stay
Time Frame: 30 days
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Goal Directed Therapy | Usual Care
Number analyzed (Participants) | 23 | 25
hours | 30.3 [24.8 to 69.8] | 42.3 [27.4 to 46.9]

6. Secondary Outcome: Hospital Length of Stay
Time Frame: 30 days
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Goal Directed Therapy | Usual Care
Number analyzed (Participants) | 23 | 25
days | 10.8 [9.3 to 19.9] | 9.0 [8.0 to 12.1]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Goal Directed Therapy | Usual Care
All-Cause Mortality (participants affected / at risk) | 2/23 | 1/25
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/25
Other Adverse Events (participants affected / at risk) | 0/23 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/55/NCT02864355/Prot_SAP_000.pdf